CLINICAL TRIAL: NCT01027884
Title: A Phase III Double-Blind, Randomised, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of Idebenone in 10-18 Year Old Patients With Duchenne Muscular Dystrophy
Brief Title: Phase III Study of Idebenone in Duchenne Muscular Dystrophy (DMD)
Acronym: DELOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-III-003
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Muscular Dystrophy, Duchenne; Ambulatory Care
Keywords: Idebenone; Duchenne Muscular Dystrophy (DMD); Respiratory function; Ambulatory and non-ambulatory patients; Subjects not using glucocorticoids
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Respiratory Aspiration | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 900 mg/day
  Interventions: Drug: Placebo
- Idebenone (Experimental): Idebenone 900 mg/day
  Interventions: Drug: Idebenone

INTERVENTIONS:
Drug: Placebo — Placebo (900 mg/day) 2 tabl (150 mg each) x 3 times orally with meals
  Arms: Placebo
Drug: Idebenone — Idebenone (900 mg/day) 2 tabl (150 mg each) x 3 times orally with meals
  Other Names: CATENA®; RAXONE®
  Arms: Idebenone

SUMMARY:
The aim of this Phase III study was to assess the efficacy of idebenone on pulmonary function, motor function, muscle strength and quality of life in patients with DMD. Furthermore, the safety and tolerability of idebenone was assessed.

DETAILED DESCRIPTION:
This study was a Phase III, multicenter, randomized, double-blind, placebo-controlled efficacy and safety study. DMD patients (ambulatory and non-ambulatory) at age 10-18 years were enrolled at sites in Europe and North America. Study subjects were randomized in a 1:1 ratio to receive either idebenone (900 mg/day) or placebo 3 times a day with meals for 52 weeks. The primary endpoint was the difference between Catena®/Raxone® and placebo in the change from Baseline to week 52 in Peak Expiratory Flow (PEF as percent predicted, PEF%p, a measure of respiratory muscle strength) as measured by hospital-based spirometry. PEF was also measured by the patient at home using the hand-held ASMA-1 device (secondary endpoint). Other respiratory endpoints included Forced Expiratory Volume in 1 second (as percent predicted, FEV1%p, an additional measure of respiratory muscle strength) and Forced Vital Capacity (as percent predicted, FVC%p, a measure of restrictive lung disease predictive of morbidity and mortality in DMD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 10 - 18 years of age at Baseline.
2. Signed and dated informed consent.
3. Documented diagnosis of DMD or severe dystrophinopathy and clinical features consistent of typical DMD at diagnosis (i.e. documented delayed motor skills and muscle weakness by age 5 years). DMD should be confirmed by mutation analysis in the dystrophin gene or by substantially reduced levels of dystrophin protein (i.e. absent or <5% of normal) on Western blot or immunostain.
4. Ability to provide reliable and reproducible repeat PEF within 15% of the first assessment (i.e. Baseline vs. Screening).
5. Patients assessed by the investigator as willing and able to comply with the requirements of the study, possess the required cognitive abilities and are able to swallow study medication.

Exclusion Criteria:

1. Patients dependent on assisted ventilation at Screening and/or Baseline (defined as non-invasive nocturnal ventilation, daytime non-invasive ventilation or continuous invasive ventilation).
2. Patients with documented DMD-related hypoventilation for which assisted ventilation is needed according to current standard of care guidelines (e.g. FVC< 30%) or is required in the opinion of the Investigator.
3. Patients with a percent predicted PEF > 80% at Baseline.
4. Patients unable to form a mouth seal to allow precise respiratory flow measurements and mouth pressures.
5. Symptomatic heart failure (high probability of death within one year of Baseline) and/or symptomatic ventricular arrhythmias.
6. Participation in the previous Phase II or Phase II Extension study (SNT-II-001 or SNT-II-001-E) for idebenone.
7. Participation in any other therapeutic trial and/or intake of any investigational drug within 90 days prior to Baseline.
8. Use of carnitine, creatine, glutamine, oxatomide, or any herbal medicines within 30 days prior to Baseline.
9. Use of coenzyme Q10 or vitamin E (if taken at a dose of 5 times above the daily physiological requirement) within 30 days prior to Baseline.
10. Any previous use of idebenone.
11. Any concomitant medication with a depressive or stimulating effect on respiration or the respiratory tract.
12. Planned or expected spinal fixation surgery during the study period (as judged by the investigator).
13. Asthma, bronchitis/COPD, bronchiectasis, emphysema, pneumonia or the presence of any other non-DMD respiratory illness that affects PEF.
14. Chronic use of beta-2 agonists or any use of other bronchodilating medication (e.g. inhaled steroids, sympathomimetics, anticholinergics).

    Please note: Chronic use if defined as a daily intake for more than 14 days.
15. Moderate or severe hepatic impairment or severe renal impairment.
16. Prior or ongoing medical condition or laboratory abnormality that in the Investigator's opinion could adversely affect the safety of the subject.

    Please note: Patients who suffer from a severe, unstable condition including (but not limited to) cancer, auto-immune diseases, haematological diseases, metabolic disorders or immunodeficiencies, and who are at risk of an aggravation unrelated to the study condition, can only be included in the study if accepted in writing by the Sponsor's Medical Monitor.
17. Relevant history of or current drug or alcohol abuse or use of any tobacco/marijuana products/smoking
18. Known individual hypersensitivity to idebenone or to any of the ingredients/excipients of the study medication
19. Systemic glucocorticoid therapy

    1. Chronic use of systemic glucocorticoid therapy for DMD related conditions within 12 months of Baseline (the "12 month non-use period")
    2. More than 2 rounds of acute systemic glucocorticoid burst therapy (of ≤2 week duration) for non-DMD related conditions within the 12 month non-use period
    3. Use of any round of systemic glucocorticoid burst therapy of longer than 2 weeks duration within the 12 month non-use period
    4. Use of systemic glucocorticoid burst therapy less than 8 weeks prior to baseline

Ages: 10 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Gunnar Buyse, MD, PhD., Principal Investigator — University Hospitals Leuven, B-3000, Belgium; Dr. Ulrike Schara, MD, PhD, Principal Investigator — Universitätsklinikum Essen, D-45122 Essen, Germany; Ass. Prof. Jan Verschuuren, MD, PhD, Principal Investigator — Leiden University Medical Center (LUMC), 2300 RC Leiden, the Netherlands; Dr. Pierre-Yves Jeannet, Médecin Associé, MER, Principal Investigator — Unité de Neuropédiatrie, CHUV - BH11, 1011 Lausanne-CH, Switzerland; Prof. Thomas Voit, MD, PhD, Principal Investigator — Université Pierre et Marie curie VI - Institut de Myologie - groupe hospitalier Pitié Salpétrière - 47/83 boulevard de l'hôpital, 75651 Paris Cedex 13, France; Prof. Thomas Sejersen, MD, PhD, Principal Investigator — Astrid Lindgrens Barnsjukhus- Karolinska Universitetssjukhuset, SE-17176 Stockholm, Sweden; Dr. Günther Bernert, Prim. Univ. Doz., Principal Investigator — Vorstand der Abteilung für Kinder- und Jugendheilkunde, Gottfried v. Preyer'sches Kinderspital, 1100 Wien, Austria; Gihan Tennekoon, MD, Principal Investigator — Division of Neurology - The Children's Hospital of Philadelphia - 34th Street and Civic Center Blvd, Philadelphia, PA 19104-1771, USA; Jean-Marie Cuisset, MD, Principal Investigator — Hôpital Roger Salengro, CHRU, Service de neurologie infantile, Lille, France; Susan Iannaccone, MD, Principal Investigator — University of Texas Southwestern Medical Center, TX, USA; Susan Sparks, MD, Principal Investigator — The Charlotte-Mecklenburg Hospital Authority, Charlotte, NC, USA; Janbernd Kirschner, MD, Principal Investigator — Universitätsklinik Freiburg Zentrum für Kinderheilkunde und Jugendmedizin; Maria Grazia Nadia D'Angelo, MD, Principal Investigator — Fondazione IRCCS "Eugenio Medea"; Ksenija Gorni, MD, Principal Investigator — Azienda Ospedaliera Niguarda Ca'Granda Centro Clinico Nemo; Bryan W. Burnette, MD, Principal Investigator — Monroe Carell Jr. Children's Hospital at Vanderbilt; Barry Byrne, MD, Principal Investigator — University of Florida; Michele Yang, MD, Principal Investigator — Children's Hospital Colorado; Susan Apkon, MD, Principal Investigator — Seattle Children's Hospital; Ericka Simpson, MD, Principal Investigator — Methodist Neurological Institute, Houston; Craig McDonald, MD, Principal Investigator — University of California, Davis; Luisa Politano, MD, Principal Investigator — Azienda Ospedaliera Universitaria della Seconda Università degli Studi di Napoli; Ana Camacho Salas, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Juan Jesus Vilchez, MD, Principal Investigator — Hospital Universitari y Politècnic La Fe de Valencia
Locations (23):
- United States (9):
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Carolinas Medical Center, Neurosciences and Spine Institute, Charlotte, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Monroe Carell, Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Methodist Neurological Institute, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Dr. Günther Bernert, Prim. Univ. Doz., Vienna, Austria
- University Hospitals Leuven- Children Hospital, Leuven, Belgium
- France (2):
  - Hôpital Roger Salengro, CHRU Lille, Lille
  - Prof. Thomas Voit , MD, PhD, Paris
- Germany (2):
  - Universitätsklinikum Essen, Zentrum für Kinderheikunde, Essen
  - Universitätsklinik Freiburg Zentrum für Kinderheilkunde und Jugendmedizin, Freiburg im Breisgau
- Italy (3):
  - Fondazione IRCCS "Eugenio Medea", Bosisio Parini, Lecco
  - Azienda Ospedaliera Niguarda Ca' Granda Centro Clinico Nemo, Milan
  - Azienda Ospedaliera Universitaria della Seconda Università degli Studi di Napoli, Napoli
- Ass. Prof. Jan Verschuuren , MD, PhD, Leiden, P.O. Box 9600, Netherlands
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia
- Prof. Thomas Sejersen, MD, PhD, Stockholm, Sweden
- CHUV Lausanne Neuropediatrie, Lausanne, Switzerland

REFERENCES:
- [Result] Buyse GM, Voit T, Schara U, Straathof CSM, D'Angelo MG, Bernert G, Cuisset JM, Finkel RS, Goemans N, McDonald CM, Rummey C, Meier T; DELOS Study Group. Efficacy of idebenone on respiratory function in patients with Duchenne muscular dystrophy not using glucocorticoids (DELOS): a double-blind randomised placebo-controlled phase 3 trial. Lancet. 2015 May 2;385(9979):1748-1757. doi: 10.1016/S0140-6736(15)60025-3. Epub 2015 Apr 20. PMID 25907158
- [Derived] Meier T, Rummey C, Leinonen M, Spagnolo P, Mayer OH, Buyse GM; DELOS Study Group. Characterization of pulmonary function in 10-18 year old patients with Duchenne muscular dystrophy. Neuromuscul Disord. 2017 Apr;27(4):307-314. doi: 10.1016/j.nmd.2016.12.014. Epub 2017 Jan 6. PMID 28189481
- See also: Related Info — http://www.santhera.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting centres were in Belgium, Germany, the Netherlands, Switzerland, France, Sweden, Austria, Italy, Spain, and the USA. Patients were enrolled between July 27, 2009 (study start date), and Dec 14, 2012; the study end date (last patient completed the study) was Jan 14, 2014.
Pre-assignment Details: 65 patients were randomly assigned and two patients were allocated to the same treatment as their randomly assigned siblings. One patient never took study medication, resulting in 66 patients who were treated and included in the safety population (34 in the placebo group and 32 in the idebenone group).
Groups:
- Placebo: Two matching placebo tablets were taken three times a day with meals
- Idebenone: Two150 mg tablets were taken three times a day with meals (total dose 900 mg daily).
Period: Overall Study
Arm/Group | Placebo | Idebenone
Started | 34 | 32
Completed | 30 | 25
Not Completed | 4 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Non-compliance | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Spinal fixation surgery | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Idebenone | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 15 (2.5) | 13.5 (2.7) | 14.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Predicted Peak Expiratory Flow (PEF) at Week 52
Description: Change from Baseline in Percent Predicted Peak Expiratory Flow (PEF) at Week 52
Time Frame: Baseline and Week 52
Population: This analysis was performed on the ITT population(n=64). This population included all randomized patients who received at least one dose of the study medication and provided at least one post-Baseline assessment. It excluded siblings who had been allocated to the same study treatment as a randomized sibling.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 33 | 31
percentage | -8.84 [-12.73 to -4.95] | -2.57 [-6.68 to 1.54]

2. Secondary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 52
Description: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 52
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of Predicted FVC
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 33 | 31
percentage of Predicted FVC | -8.95 [-11.47 to -6.42] | -5.67 [-8.36 to -2.99]

3. Secondary Outcome: Change From Baseline to Week 52 in Muscle Strength
Description: The change from Baseline to Week 52 in muscle strength as measured by Hand-Held Myometry (HHM) was performed following standardized procedures. As almost all patients were non-ambulatory, only analyses of upper limb muscle strength were performed. Results for elbow flexors and for elbow extensors are reported below.The highest value of 3 consecutive measurements with an interval of at least 10 seconds were recorded.
  The HHM was measured using MicroFET2, a digital hand held muscle tester. The selected unit of measure was Newtons (N).
Time Frame: Baseline and Week 52
Population: The number of patients (N) in each treatment group is the number of patients with baseline assessments
Measure: Mean (95% Confidence Interval); unit: Newtons
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 27 | 25
Newtons
  Elbow Flexors | 0.13 [-4.16 to 4.41] | -2.32 [-6.73 to 2.09]
  Elbow Extensors | 1.32 [-2.53 to 5.18] | 0.26 [-3.95 to 4.46]

4. Secondary Outcome: Change From Baseline to Week 52 in Quality of Life Assessed by PedsQL™ Paediatric Quality of Life Inventory
Description: PedsQL Quality of Life Inventory contains paediatric HRQOL measurements: Physical, Emotional,Social and School Functioning.
  Item Scaling:
  5-point Likert scale from 0 (Never) to 4 (Almost always). 3-point scale: 0 (Not at all), 2 (Sometimes) and 4 (A lot) for the Young Child (ages 5-7).
  Scores are transformed on a scale from 0 to 100 ( 0=100, 1=75, 2=50, 3=25, 4=0) Total Score: Sum of all the items over the number of items answered on all the Scales.
  The values reported below are overall scores on Paediatric Quality of Life Inventory in Child/Teen Report. These scores were obtained by averaging scores for all the described subscales. The overall scores range between 0-100 with 0 = worst outcome and 100= best outcome
Time Frame: Baseline and Week 52
Population: The number of patients (N) in each treatment group is the number of patients with Baseline assessments.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 33 | 30
units on a scale | 2.46 [-1.77 to 6.69] | -1.34 [-5.99 to 3.31]

5. Secondary Outcome: Percentage of Patients Reporting Adverse Events
Time Frame: 52 Weeks
Measure: Number; unit: percentage of patients reporting AEs
Arm/Group | Placebo | Idebenone
Number analyzed (Participants) | 34 | 32
percentage of patients reporting AEs | 94.1 | 93.8

ADVERSE EVENTS:
Arm/Group | Placebo | Idebenone
Serious Adverse Events (participants affected / at risk) | 5/34 | 2/32
Other Adverse Events (participants affected / at risk) | 32/34 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | Idebenone (N=32)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmunary microemboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Psychiatric disorders) | 0 | 1
Vomitig (Gastrointestinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | Idebenone (N=32)
Left ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Electrocardiogram abnormal (Cardiac disorders) | 1 (1) | 2 (3)
Blood phosporus increased (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 7 (15) | 6 (13)
Pyrexia (General disorders) | 3 (4) | 5 (6)
Influenza like illness (General disorders) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 8 (10)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 9 (11) | 8 (12)
Upper respiratory tract infection (Infections and infestations) | 6 (10) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 6 (7)
Rhinitis (Infections and infestations) | 6 (8) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No